CLINICAL TRIAL: NCT01015430
Title: A Randomized, Double-blind, Placebo-controlled, Pharmacokinetic, Safety and Tolerability, and Exploratory Efficacy and Pharmacodynamic Effects Study of RO4917523 in Adult Patients With Fragile X Syndrome.
Brief Title: A Study With RO4917523 in Patients With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP22578
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Placebo (for RO4917523 ascending doses) (Placebo Comparator)
  Interventions: Drug: Placebo (for RO4917523 ascending doses); Drug: Placebo (for RO4917523 fixed dose)
- Placebo (for RO4917523 fixed dose) (Placebo Comparator)
  Interventions: Drug: Placebo (for RO4917523 ascending doses); Drug: Placebo (for RO4917523 fixed dose)
- RO4917523 ascending doses (Experimental)
  Interventions: Drug: RO4917523
- RO4917523 fixed dose (Experimental)
  Interventions: Drug: RO4917523

INTERVENTIONS:
Drug: Placebo (for RO4917523 ascending doses) — Placebo daily po
  Arms: Placebo (for RO4917523 ascending doses); Placebo (for RO4917523 fixed dose)
Drug: Placebo (for RO4917523 fixed dose) — Placebo daily po
  Arms: Placebo (for RO4917523 ascending doses); Placebo (for RO4917523 fixed dose)
Drug: RO4917523 — RO4917523 ascending doses daily po
  Arms: RO4917523 ascending doses
Drug: RO4917523 — RO4917523 fixed dose daily po
  Arms: RO4917523 fixed dose

SUMMARY:
This randomized, double-blind multiple ascending dose study will evaluate the safety and tolerability, pharmacokinetics and efficacy of RO4917523 in patients with Fragile X Syndrome. The patients will be randomized to receive either active drug or placebo. The anticipated time on study treatment is 6 weeks. The target sample size is <100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 to 50 years of age
* Fragile X Syndrome
* IQ less than 75
* Reliable caregiver

Exclusion Criteria:

* Current psychosis or presumption of psychosis
* History of suicidal behavior or considered a high suicidal risk
* Severe self-injurious behavior
* Any unstable medical condition other than Fragile X Syndrome (e.g. hypertension, diabetes)
* Current seizure disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety, Tolerability and Pharmacokinetics: AEs, laboratory parameters | AEs throughout study; laboratory assessments: days 1, 8, 15, 29, 43

SECONDARY OUTCOMES:
Efficacy: Behavior and cognition assessments | Every 2 weeks throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - Sacramento, California
  - Decatur, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Nashville, Tennessee